CLINICAL TRIAL: NCT05541601
Title: Prospective Cohort for Early Detection of Liver Cancer
Acronym: Pearl
Status: Recruiting | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Cancer Research UK (Other); Roche Diagnostic Ltd. (Industry); OncImmune Ltd (Unknown); Perspectum (Industry); University of Nottingham (Other); Glasgow Caledonian University (Other)
Responsible Party: Sponsor
Other Study IDs: Pearl
Record Dates: First submitted 2022-08-01; First posted 2022-09-15 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Cirrhosis; Hepatocellular Carcinoma
MeSH Terms: conditions — Fibrosis; Carcinoma, Hepatocellular | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pearl Cohort: All 3000 patients recruited to the Pearl study
  Interventions: Other: Blood and Urine samples

INTERVENTIONS:
Other: Blood and Urine samples — The samples will be used to identify a range of tests (including genetic, protein and other biomarkers), which along with the clinical data will hopefully identify those most at risk of developing HCC, and to identify HCC at the earliest possible time points.

SUMMARY:
This study aims to recruit 3000 people with liver cirrhosis into a Prospective cohort for early detection of Liver cancer - the Pearl cohort. The study team believe that using a combination of novel tests may improve the detection of early Hepatocellular Carcinoma (HCC).

DETAILED DESCRIPTION:
During a four-year follow-up period, around 100 Pearl patients are expected to be diagnosed with HCC. Blood, urine, clinical and imaging data will be collected over the follow up period. The samples will be used to identify a range of tests (including genetic, protein and other biomarkers), which along with the clinical data will hopefully identify those most at risk of developing HCC, and to identify HCC at the earliest possible time points.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of all genders, age >18 years
2. Participant is willing and able to give informed consent for participation in the study.
3. Evidence of cirrhosis CP A or B (as defined below, cirrhosis ever diagnosed), with an underlying aetiology of at least one of the following: chronic Hepatitis B Virus (HBV) infection, chronic Hepatitis C Virus (HCV) infection, alcoholic liver disease, non-alcoholic fatty liver disease or haemochromatosis

Cirrhosis Diagnosis Definition

1. Histological assessment (Ishak stage 5 or 6) or
2. At least one of the following:

i. Validated non-invasive marker of fibrosis including fibroscan, AST to Platelet Ratio Index (APRI) score >2 or Enhanced Liver Fibrosis (ELF) score >10.48 or Fibrotest score >0.73. Fibroscan readings should be assessed by aetiology as below:

* HBV: >=10 kPa
* HCV: >=14.5 kPa
* Alcoholic Liver Disease (ALD): >=19.5 kPa
* Non-alcoholic fatty liver disease (NAFLD): >=15 kPa
* Haemochromatosis: >=12kPa ii. Evidence of varices at endoscopy or imaging in the context of a patent portal vein iii. Definitive radiological evidence of cirrhosis (i.e. nodularity of liver and splenomegaly on Ultrasound/CT)

Exclusion Criteria:

1. Diagnosis of current OR historical hepatocellular carcinoma
2. Liver transplant recipients or patients on active listing for liver transplantation
3. Child-Pugh C cirrhosis
4. In the view of the clinician, if the patient has a co-morbidity likely to lead to death within the following 12 months
5. In the view of the clinician, if the patient was not thought to be suitable for HCC surveillance

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with Child-Pugh (CP) A or B cirrhosis with no current or historical diagnosis of HCC. Diagnosis of cirrhosis can be based on, laboratory, imaging or histology criteria (e.g. the latter including Ishak stage >=5). Participants can be recruited to other interventional studies for treatment of cirrhosis or prevention of HCC prior to or during participation in the Pearl study.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-02-23 (Actual); Primary Completion 2037-07 (Estimated); Study Completion 2037-07 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of novel diagnostic approaches for the early diagnosis of HCC in enrolled patients who are diagnosed with HCC by conventional approaches. | When 50 cases of HCC have accumulated through to study completion; up to 5 years
  Diagnostic approaches to be tested will include:
  1. detection of epigenetic (e.g. methylation profiling) and genetic mutations, and copy number variations in circulating tumour DNA;
  2. multiparametric MRI liver imaging including MR biomarkers of inflammation, fibrosis, fat and iron content;
  3. host genetic makeup (relevant variants identified through Genome Wide Association Studies);
  4. detection of autoantibodies to tumour associated antigens;
  5. epitope mapping of circulating antibody repertoire using random peptide libraries;
  6. protein biomarkers including the L3 isoform of alphafetoprotein, and des-gammacarboxy- prothrombin;
  7. proteomic and metabolomic profiling, including steroid metabolic signatures in urine.
Specificity of novel diagnostic approaches for the early diagnosis of HCC in enrolled patients who are diagnosed with HCC by conventional approaches. | When 50 cases of HCC have accumulated through to study completion; up to 5 years
  Diagnostic approaches to be tested will include:
  1. detection of epigenetic (e.g. methylation profiling) and genetic mutations, and copy number variations in circulating tumour DNA;
  2. multiparametric MRI liver imaging including MR biomarkers of inflammation, fibrosis, fat and iron content;
  3. host genetic makeup (relevant variants identified through Genome Wide Association Studies);
  4. detection of autoantibodies to tumour associated antigens;
  5. epitope mapping of circulating antibody repertoire using random peptide libraries;
  6. protein biomarkers including the L3 isoform of alphafetoprotein, and des-gammacarboxy- prothrombin;
  7. proteomic and metabolomic profiling, including steroid metabolic signatures in urine.
Positive/Negative predictive values of novel diagnostic approaches for the early diagnosis of HCC in enrolled patients who are diagnosed with HCC by conventional approaches. | When 50 cases of HCC have accumulated through to study completion; up to 5 years
  Diagnostic approaches to be tested will include:
  1. detection of epigenetic (e.g. methylation profiling) and genetic mutations, and copy number variations in circulating tumour DNA;
  2. multiparametric MRI liver imaging including MR biomarkers of inflammation, fibrosis, fat and iron content;
  3. host genetic makeup (relevant variants identified through Genome Wide Association Studies);
  4. detection of autoantibodies to tumour associated antigens;
  5. epitope mapping of circulating antibody repertoire using random peptide libraries;
  6. protein biomarkers including the L3 isoform of alphafetoprotein, and des-gammacarboxy- prothrombin;
  7. proteomic and metabolomic profiling, including steroid metabolic signatures in urine.

SECONDARY OUTCOMES:
To develop models that can be used to "risk-stratify" cirrhosis patients according to their future risk of HCC | Throughout study to completion; 5 years
  The Harrell's Concordance Index (C-index) will be calculated for each biomarker/model of interest. The minimum and maximum C-index scores are 0 and 1, respectively, where the higher the score the better the biomarker/model is at identifying HCC risk. C-index values indicate the degree to which individuals who develop HCC have a higher risk score than those who do not. C-index values will be adapted to incorporate non-HCC mortality as a competing risk. The C-index value will be used to identify the biomarkers/models with the best discriminative ability.
To better understand the incidence of HCC in a UK population stratified by underlying cirrhosis aetiology | At 1, 3 and 5 year post- baseline.
  Cumulative incidence of HCC according to cirrhosis aetiology

CONTACTS AND LOCATIONS:
Overall Officials: Ellie Barnes, Principal Investigator — University of Oxford
Locations (1):
- Hepatology Clinical Trial Unit, John Radcliffe Hospital, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Derived] Khanna K, Barnes E, Benselin J, Culver E, Irving W, Innes H, Pavlides M, Consortium D. Prospective cohort for early detection of liver cancer (Pearl): a study protocol. BMJ Open. 2024 Oct 1;14(10):e085541. doi: 10.1136/bmjopen-2024-085541. PMID 39353693
- See also: DeLIVER Project Website — https://deliver.cancer.ox.ac.uk/